CLINICAL TRIAL: NCT02590666
Title: Comparative Study of Endometrial Polypectomy Performed With Bipolar Electrode Versapoint vs Microscissors or Graspers
Brief Title: Endometrial Polypectomy Performed With Bipolar Electrode Versapoint vs Microscissors or Graspers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PolypectomyCA
Record Dates: First submitted 2015-10-25; First posted 2015-10-29 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Endometrial Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bipolar electrode (Experimental): Polyps resection with bipolar electrode
  Interventions: Procedure: Bipolar Polypectomy; Device: Bipolar electrode
- Microscissors or graspers (Active Comparator): Polyps resection with microscissors or graspers
  Interventions: Procedure: Mechanical Polypectomy; Device: Microscissors or graspers

INTERVENTIONS:
Procedure: Bipolar Polypectomy — Polyps resection with bipolar electrode
  Arms: Bipolar electrode
Procedure: Mechanical Polypectomy — Polyps resection with microscissors or graspers
  Arms: Microscissors or graspers
Device: Bipolar electrode — Bipolar electrode used to performs polypectomy
  Arms: Bipolar electrode
Device: Microscissors or graspers — Mechanical instruments used to performs polypectomy
  Arms: Microscissors or graspers

SUMMARY:
Hysteroscopy today is considered the gold standard for the diagnosis and treatment of endometrial polyps. Several hysteroscopic systems to resect endometrial polyps are currently available. Among Others bipolar systems and microscissors or graspers, both of theme make part of routine clinical practice and are universally accepted.

The aim of the study is to compare the efficacy of bipolar resection energy polypectomy versus microscissors or graspers These procedures assume a lower cost and are associated with a lower surgical risk due to their realization without anesthesia .

Hypothesis: Resection of polyps outpatient laser diode has a similar or superior to that of the bipolar electrode tolerability. The diode laser is a viable , quick , simple technique with a high percentage of resection and high degree of satisfaction of patients

ELIGIBILITY:
Inclusion Criteria:

* The patient must be informed about the study, and sign the informed consent

Exclusion Criteria:

* Positive Pap smear test
* Pregnancy
* Uterine malignancy
* Abnormal uterine bleeding

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
To assess the tolerability of polypectomy using a validated visual analogue pain scale | we measure pain after resection of endometrial polyps, with 5 minutes for the patient thinks

OTHER OUTCOMES:
Assess the recurrence of polyps after 3 months of resection (another hysteroscopy). | 3 months after resection of the polyp, repeat hysteroscopy to assess recurrence